CLINICAL TRIAL: NCT04155229
Title: Effect of Default Electronic Health Record Settings on Clinician Opioid Prescribing Patterns in Emergency Departments
Brief Title: EMR Defaults to Nudge Opioid Prescribing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: EMRdefaults
Record Dates: First submitted 2019-10-28; First posted 2019-11-07 (Actual); Last update posted 2019-11-07 (Actual); Status verified 2019-11

CONDITIONS: Pain, Acute; Opioid Use, Unspecified
MeSH Terms: conditions — Acute Pain | interventions — Acetaminophen; Hydrocodone; Oxycodone; oxycodone-acetaminophen

STUDY DESIGN:
Intervention Model Description: Each of two sites underwent block randomization of four treatment assignments.
Masking Description: The investigators did not mask the changes to the electronic medical record, but note that they also did not announce them.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Null setting, forced entry (Experimental): Each arm sets the default quantity (preset quantity) embedded in the electronic medical record for study opioids.
  This arm has a default setting for opioid quantity set at -blank-. This setting required the prescriber to enter a quantity in order to write a prescription.
  Interventions: Other: Default settings for opioid prescriptions (acetaminophen/hydrocodone, oxycodone, acetaminophen/oxycodone)
- 5 tablet default (Experimental): Each arm sets the default quantity (preset quantity) embedded in the electronic medical record for study opioids.
  This arm has a default setting for opioid quantity set at 5.
  Interventions: Other: Default settings for opioid prescriptions (acetaminophen/hydrocodone, oxycodone, acetaminophen/oxycodone)
- 10 tablet default (Experimental): Each arm sets the default quantity (preset quantity) embedded in the electronic medical record for study opioids.
  This arm has a default setting for opioid quantity set at 10.
  Interventions: Other: Default settings for opioid prescriptions (acetaminophen/hydrocodone, oxycodone, acetaminophen/oxycodone)
- 15 tablet default (Experimental): Each arm sets the default quantity (preset quantity) embedded in the electronic medical record for study opioids.
  This arm has a default setting for opioid quantity set at 15.
  Interventions: Other: Default settings for opioid prescriptions (acetaminophen/hydrocodone, oxycodone, acetaminophen/oxycodone)
- Status quo default setting (Active Comparator): Each arm sets the default quantity (preset quantity) embedded in the electronic medical record for study opioids.
  This arm has a default setting for opioid quantity set at the status quo value for each site (20 for site 1, 12 for site 2).
  Interventions: Other: Default settings for opioid prescriptions (acetaminophen/hydrocodone, oxycodone, acetaminophen/oxycodone)

INTERVENTIONS:
Other: Default settings for opioid prescriptions (acetaminophen/hydrocodone, oxycodone, acetaminophen/oxycodone) — For each of the arms, the investigators modified the default setting for the dispense quantity of study opioids on the electronic medical record settings for discharge prescriptions.
  Study drugs include acetaminophen 325mg + hydrocodone 5mg, acetaminophen 325mg + hydrocodone 7.5mg, acetaminophen 325mg + hydrocodone 10mg, oxycodone 5mg, acetaminophen 325mg + oxycodone 5mg, acetaminophen 325mg + oxycodone 10mg.

SUMMARY:
The investigators conducted a prospective, block-randomized study to determine whether and to what extent changes in the default settings in the electronic medical record (EMR) affect opioid prescriptions for patients discharged from emergency departments (EDs).

DETAILED DESCRIPTION:
In two large, urban emergency departments, we randomly altered the pre-populated dispense quantities of discharge prescriptions for commonly-prescribed opioids over a series of five 4-week blocks. These changes were made without announcement, and providers were not informed of the study itself.

ELIGIBILITY:
Inclusion Criteria:

* Discharge prescription from emergency for study drug: hydrocodone/acetaminophen, oxycodone, or oxycodone/acetaminophen.

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2016-10-03 (Actual); Primary Completion 2017-09-03 (Actual); Study Completion 2017-09-03 (Actual)

PRIMARY OUTCOMES:
Dispense quantity of prescribed opioids | Through study completion, approximately 340 days
  The dispense quantity of prescribed study drugs was collected from the electronic medical record at each site. The mean and median quantities per prescription according to each study arm were compared.

SECONDARY OUTCOMES:
Proportion ≤12 | Through study completion, approximately 340 days
  The dispense quantity of study drugs was collected from the electronic medical record at each site. The proportion of prescriptions at 12 or fewer tablets was compared across study arms.
Proportion at default setting | Through study completion, approximately 340 days
  The dispense quantity of study drugs was collected from the electronic medical record at each site. The proportion of prescriptions written for the given default setting was compared across treatment arms.

CONTACTS AND LOCATIONS:
Overall Officials: Juan Carlos Montoy, MD, PhD, Principal Investigator — University of California, San Francisco

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Montoy JCC, Coralic Z, Herring AA, Clattenburg EJ, Raven MC. Association of Default Electronic Medical Record Settings With Health Care Professional Patterns of Opioid Prescribing in Emergency Departments: A Randomized Quality Improvement Study. JAMA Intern Med. 2020 Apr 1;180(4):487-493. doi: 10.1001/jamainternmed.2019.6544. PMID 31961377